CLINICAL TRIAL: NCT06603350
Title: The Effect of Perioperative Factors on Postoperative Outcomes in Patients Undergoing Lung Transplantation: a Prospective Observational Study
Brief Title: The Effect of Perioperative Factors on Postoperative Outcomes After Lung Transplantation
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0764
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Complications After Lung Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Peripheral blood serum at 5 timepoints，before ansethesia induction, at the end of surgery, 24h after surgery, 48h after surgery and 72h after surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intenvention — No intenvention

SUMMARY:
1. Evaluate the influence of perioperative factors on postoperative outcomes in patients undergoing lung transplantation patients.
2. To evaluate the feasibility of using pulmonary ultrasound to identify lung complications such as atelectasis and pulmonary edema after lung transplantation
3. Observe the changes of perioperative inflammation and immune indexes after lung transplantation

ELIGIBILITY:
Inclusion Criteria:

Prosedure of lung transplantation, Aged more than 18 years old

Exclusion Criteria:

Secondary lung transplantation, multiple organ transplantation, refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria are adult patients undergoing lung transplantation Those undergoing retransplantation,multiple organ transplantation or refusal to participate will be excluded.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-28 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | 3 days after surgery
  Incidence of atelectasis and primary graft dysfunction(PGD) detcted by lung ultrasound
Mortality | 1 year after surgery
  Survival rate after lung transplantation

SECONDARY OUTCOMES:
Inflammatory index IL-6 | 3 days after after surgery
  Variation of perioperative inflammatory index IL-6

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No